CLINICAL TRIAL: NCT01976533
Title: Eisenmenger Syndrome in the Nordic Countries: Advanced Treatment and Mortality 1977-2012
Brief Title: Eisenmenger Syndrome in the Nordic Countries
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Lund University Hospital (Other); Rikshospitalet University Hospital (Other); Hospital for Children and Adolescents, Finland (Other); Actelion (Industry)
Responsible Party: Principal Investigator, Cristel Sørensen, MD, Rigshospitalet, Denmark
Other Study IDs: 3-3013-144/1/
Record Dates: First submitted 2013-10-29; First posted 2013-11-06 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Eisenmenger Syndrome
MeSH Terms: conditions — Eisenmenger Complex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Advanced therapy, Heart-lung transplantation, dead

SUMMARY:
This is a historical cohort study with retrospective collection of data comprising all Nordic patient's diagnosed with Eisenmengers syndrome in the period 1977 through 2011. The goal is to determine prognostic factors for mortality and morbidity.

DETAILED DESCRIPTION:
The following variables are obtained from national registries for each individual fulfilling the inclusion criteria:

* Personal data: Gender, day of birth, vital status (dead/alive), date of death, cause of death, all cause hospitalization days
* Specific cardiac malformation diagnosis
* Heart-lung transplantation.
* Social data: Highest educational level, marital status, employment status (Denmark only)

Primary endpoints

* Incidence and prevalence of Eisenmenger Syndrome
* All-cause mortality
* All-cause morbidity (hospitalization for any cause)
* Heart-lung transplantation
* Advanced treatment
* Mortality with AT
* Highest educational level
* Personal income
* Marital status
* Job status

ELIGIBILITY:
Inclusion Criteria:

* Eisenmenger syndrome

Exclusion Criteria:

-

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Nordic patients with Eisnemnger syndrome
Sampling Method: Probability Sample
Enrollment: 714 (Actual)
Dates: Start 2012-10; Primary Completion 2015-12 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Lars Soendergaard, MD, DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (4):
- Dept. Cardiology B, Rigshospitalet, Copenhagen, Denmark
- Centers for Adult Congenital Heart Disease, Various, Finland
- Centers for Adult Congenital Heart Disease, Various, Norway
- Centers for adult congenital heart disease, Various, Sweden